CLINICAL TRIAL: NCT01592656
Title: Long-term Effects of Non-invasive Ventilation in Hypercapnic COPD Patients.
Brief Title: Long-term Effects of Non-invasive Ventilation in Hypercapnic Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of budget
Sponsor: FLUIDDA nv (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLUI-2010-68
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; GOLD stages II, III and IV; Computed Tomography scan; Functional Respiratory Imaging; Non-Invasive Ventilation; Arterial Blood Gas; Hypercapnic; Health Related Quality of Life; Lung compliance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypercapnia | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-invasive ventilation (NIV) (Active Comparator): 30 patients will receive NIV during 6 months = group 1
  Interventions: Radiation: Functional Respiratory Imaging; Other: Lung compliance measurement; Device: Non-invasive ventilation (Respironics)
- Control group (Placebo Comparator): 10 patients will act as control group, they will not be treated with NIV = group 2
  Interventions: Radiation: Functional Respiratory Imaging; Other: Lung compliance measurement

INTERVENTIONS:
Radiation: Functional Respiratory Imaging — CT-scan of thorax. At baseline, after 1 month and after 6 months.
Other: Lung compliance measurement — At baseline
Device: Non-invasive ventilation (Respironics) — Long-term non-invasive ventilation, starting at baseline until 6 months. At baseline the patients should have persisting hypercapnia (pCO2 > 45 mmHg) under optimal conservative treatment other than NIV. The patients can be hospitalised or being treated at home at inclusion.
  Other Names: Trilogy device (Respironics)
  Arms: Non-invasive ventilation (NIV)

SUMMARY:
In this multicenter study the comparison of the mass flow distribution and redistribution versus the relative blood flow per lobe (as a surrogate for Ventilation/ Perfusion (V/Q) matching) with functional respiratory imaging (FRI) and arterial blood gas (ABG) values will be evaluated in hypercapnic Chronic Obstructive Pulmonary Disease (COPD) patients. Therefore a low dose Computed Tomography (CT) scan will be taken in a population of 30 patients with non-invasive ventilation (NIV) and in a control group of 10 patients without NIV. The CT-scan will be used for FRI.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 40 years old
* Men and women
* Written informed consent obtained
* COPD patients GOLD II, III and IV
* Persisting hypercapnia (pCO2 > 45 mmHg ) notwithstanding adequate treatment modalities (including oxygen) as proposed by the GOLD guidelines
* Stopped smoking
* Total lung capacity (TLC) > 85%

Exclusion Criteria:

* Treatment with home NIV or Continuous Positive Airway Pressure (CPAP)
* Asthma
* Restrictive lung disease
* Symptomatic or uncontrolled heart failure
* Current malignancy
* Suspected bad compliance for NIV treatment
* Pregnant women
* Not be able to speak the language of the participating center
* Received an investigational product within 4 weeks prior to inclusion in the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Changes in the distribution of the mass flow per lobe and the relative proportion of bloodvessels, as obtained from functional respiratory imaging (FRI) and arterial blood gas (ABG). | At baseline, after 1 month and after 6 months of treatment with non-invasive ventilation (NIV)
  The primary objective of this study is the comparison of the mass flow distribution and redistribution versus the relative blood flow per lobe (as a surrogate for V/Q matching) with FRI and ABG values in hypercapnic COPD patients treated with long-term NIV.

SECONDARY OUTCOMES:
Health related quality of life | At baseline, after 1 month and after 6 months
  Saint George's Respiratory Questionnaire (SGRQ) and Severe Respiratory Insufficiency (SRI) Questionnaire
Lung function tests | At baseline, after 1 month and after 6 months
  Spirometry, reversibility, plethysmography, diffusion, Maximal Inspiratory Pressure (MIP), Maximal Expiratory Pressure (MEP)
Hospital admissions | After 1 month and after 6 months
  Length and frequency of admission, severity of exacerbations, ICU admissions
Exercise tolerance | At baseline, after 1 month and after 6 months
  6 minutes walking test and oximetry measurement
Local airway volume and resistance | At baseline, after 1 month and after 6 months
  CT-scan of thorax. CT scan is performed with a low radiation protocol. These images are made to perform computational fluid dynamics on in order to obtain more information on regional lung function characteristics.
Prediction of breathing pattern | At baseline
  The tertiary objective of the study is to predict the breathing pattern (including tidal volume) during NIV when using the data of patient specific lobar compliance and regional resistance at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Backer, MD, PhD, Principal Investigator — University Hospital, Antwerp; Peter Wijkstra, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Antwerp University Hospital, Edegem, Antwerp, Belgium
- University Medical Center Groningen, Groningen, Netherlands